CLINICAL TRIAL: NCT02824276
Title: Sensory Effects of Oral Opioid Treatment in Patients With Chronic Low Back Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Robert Edwards, Associate Professor of Anesthesia, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016P000725
Record Dates: First submitted 2016-06-28; First posted 2016-07-06 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2023-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Oxycodone; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Opioid Medication (Experimental): The primary study medication will be oxycodone, with morphine sulfate immediate release (MSIR) as a backup in case of side effects
  Interventions: Drug: Oxycodone or morphine sulfate immediate release (MSIR)
- Placebo Treatment (Placebo Comparator): Placebo medications will be encapsulated in an opaque blinding capsule to ensure adequate blinding of study medications
  Interventions: Drug: Placebo Treatment

INTERVENTIONS:
Drug: Oxycodone or morphine sulfate immediate release (MSIR) — Oxycodone or morphine sulfate immediate release (MSIR)
  Other Names: Oral Opioid Medication
  Arms: Oral Opioid Medication
Drug: Placebo Treatment — Lactose (Appearance and Weight-matched placebo capsules)
  Arms: Placebo Treatment

SUMMARY:
Chronic low back pain (CLBP) afflicts up to 50 million U.S. adults and is a primary cause of disability and reduced quality of life. The prescription of opioids for chronic low back pain (CLBP) has increased substantially within the past decade in the U.S. As noted by the CDC in their recent Guideline (released in March 2016): "Opioids are commonly prescribed for pain. An estimated 20% of patients presenting to physician offices with noncancer pain symptoms or pain-related diagnoses (including acute and chronic pain) receive an opioid prescription. Interestingly, patients scoring very high on measures of psychological distress tend to be systematically excluded from RCTs, even though this subgroup of patients is highly prevalent within the chronic pain population.

This study will provide key information on individual differences in the outcomes of opioid treatment, and its findings should facilitate more effective tailoring of analgesic regimens to individual patient characteristic.

DETAILED DESCRIPTION:
Changes in pain sensitivity will be examined (i.e., OIH) among subgroups of CLBP patients prescribed oral opioid therapy.

Investigators will conduct a moderate-term, double-blind, randomized controlled trial, and use quantitative sensory testing (QST) to evaluate whether changes in pain sensitivity and pain modulation occur as a result of long-term opioid use. Investigators hypothesize that increases in pain sensitivity (i.e., OIH) and maladaptive changes in endogenous pain modulation (i.e., enhanced temporal summation of pain) will occur as a result of long-term opioid use, but that these changes will be observed predominantly among patients with high levels of negative affect and pain-related catastrophizing.

ELIGIBILITY:
Inclusion Criteria:

1. age 25-65
2. CLBP lasting for more than 6 months as the primary complaint
3. typical pain ratings ≥ 4/10 on a visual analogue scale
4. candidate for oral opioid therapy as assessed at the BWH Pain Management Center
5. able to speak and understand English.

Exclusion Criteria:

1. evidence of delirium, dementia, psychosis, or other cognitive impairment preventing completion of study procedures
2. current (i.e., active) substance use disorder (SUD)
3. past history of persistent opioid use (i.e., opioid use for more than 6 months) given that this could affect the biological systems of interest in the present study
4. history of myocardial infarction or other serious cardiovascular condition
5. current peripheral neuropathy
6. current pregnancy, or intention to become pregnant during the study
7. current intrathecal pump.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in Pain Sensitivity (Quantitative Sensory Testing) | 6 months
  Pain Sensitivity will be assessed by Quantitative Sensory testing

CONTACTS AND LOCATIONS:
Overall Officials: Robert Edwards, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No